CLINICAL TRIAL: NCT02253706
Title: Oxygen Supplementation During Bronchoscopy: High-Flow Nasal Cannula or Low-Flow Nasal Cannula
Brief Title: Oxygen Supplementation During Bronchoscopy: High Flow Versus Low Flow Oxygen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HFO-Rx1
Record Dates: First submitted 2014-09-02; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-07

CONDITIONS: Hypoxia
Keywords: bronchoscopy; hypoxia; oxygen supplementation; safety
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low flow nasal oxygen supplementation (Active Comparator): Low flow nasal oxygen supplementation as per routine standard of care(control arm)
  Interventions: Device: low flow nasal oxygen supplementation
- High flow nasal oxygen supplementation (Experimental): High-flow nasal ventilation: This will be carried out using the Precision Flow device (Opti-Flow, Auckland, New Zealand). This device is intended to add warm moisture to breathing gases from an external source. Flow rate via the nasal cannula will be kept at 50 Liters/min and fractional inspired oxygen concentration will be set at 0.35
  Interventions: Device: High flow nasal oxygen supplementation

INTERVENTIONS:
Device: High flow nasal oxygen supplementation — High-flow nasal ventilation: This will be carried out using the Precision Flow device (Opti-Flow, Auckland, New Zealand). This device is intended to add warm moisture to breathing gases from an external source. Flow rate via the nasal cannula will be kept at 50 Liters/min and fractional inspired oxygen concentration will be set at 0.35.
  Other Names: Precision Flow device (Opti-Flow, Auckland, New Zealand)
  Arms: High flow nasal oxygen supplementation
Device: low flow nasal oxygen supplementation — Low-flow nasal ventilation: This will be carried out using a regular nasal cannula fed with oxygen at flow rates from 2 to 6 liters/minute.
  Arms: Low flow nasal oxygen supplementation

SUMMARY:
In general bronchoscopy is a safe procedure with low rate of complications. Indeed, contraindications to flexible bronchoscopy are mostly relative rather than absolute. This is the case of preexisting decreased blood oxygen levels which may be present in patients requiring further bronchopulmonary investigation. To avoid the deleterious effects of oxygen drops oxygen supplementation is recommended.

The purpose of this study is to evaluate the efficiency and safety of oxygen supplementation obtained with the use of a high flow nasal cannula compared with a low flow nasal cannula during flexible bronchoscopy.

Consecutive patients referred by their treating physician for bronchoscopy will be offered to take part in the study. Those who wish to participate and give their consent will be randomly assigned into one of two treatment groups (supplemental oxygen given via low flow nasal cannula or via high flow nasal cannula).

Assignment to either treatment arm will not affect in any way the intended purpose of the bronchoscopy. All patients will be closely monitored during the procedure and 2 hours following its completion. Monitoring will be conducted, using strictly non-invasive measures.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo routine bronchoscopy for diagnostic purposes

Exclusion Criteria:

* inability to give an informed consent
* nasal deformities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Oxygen desaturation index 4% (ODI4%) | duration of bronchoscopy with an expected average duration of 30 minutes
oxygen cumulative time below 88%(OCT88%) | beginning to end of bronchoscopy procedure with an expected average duration of 30minutes

SECONDARY OUTCOMES:
number of bradycardic and tachycardic events | beginning to end of bronchoscopy with an expected averag duration of 30 minutes
change in expired end tidal carbon dioxide before and after completion of bronchoscopy | beginning to end of bronchoscopy with an expected average duration of 30 minutes
oxygen desaturation index 4% | preprocedural to 2 hours post procedure with an expected total duration of 3 hours
cumulative oxygen time 88% | pre-procedural to 2 hours post precedure with an expected total duration of 3 hours

OTHER OUTCOMES:
patient comfort during the procedure | duration of bronchoscopy procedure with an expected average duration of 30 minutes
  a numeric rating scale ranging from 1(excellent to 4(poor ) will be filled out by the patient after completion of the bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Romem, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Albertini R, Harrel JH, Moser KM. Letter: Hypoxemia during fiberoptic bronchoscopy. Chest. 1974 Jan;65(1):117-8. doi: 10.1378/chest.65.1.117. No abstract available. PMID 4809326
- [Background] Matsushima Y, Jones RL, King EG, Moysa G, Alton JD. Alterations in pulmonary mechanics and gas exchange during routine fiberoptic bronchoscopy. Chest. 1984 Aug;86(2):184-8. doi: 10.1378/chest.86.2.184. PMID 6744959
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Roca O, Masclans JR, Laborda C, Sacanell J, Serra J. High-flow nasal cannula improves oxygenation in hypoxemic respiratory failure. Intensive Care Med 2007; 33:S86
- [Background] Williams AB, Ritchie JE, Gerard C. Evaluation of a high-flow nasal oxygen delivery system: gas analysis and pharyngeal pressures. Intensive Care Med 2006; 32: S219
- [Background] Lomas C, Roca O, Alvarez A, Masclans JR. Fibroscopy in patients with hypoxemic respiratory insufficiency: Utility of the high-flow nasal cannula. Respr Med (CME) 2009; 2: 121-124
- [Background] Lucangelo U, Vassallo FG, Marras E, Ferluga M, Beziza E, Comuzzi L, Berlot G, Zin WA. High-flow nasal interface improves oxygenation in patients undergoing bronchoscopy. Crit Care Res Pract. 2012;2012:506382. doi: 10.1155/2012/506382. Epub 2012 May 20. PMID 22666567